CLINICAL TRIAL: NCT02780076
Title: Recovery of Physical Functioning, Activity Level, and Quality of Life After Hip Fracture in the Fragile Elderly
Brief Title: Recovery of Physical Functioning After Hip Fracture
Acronym: HIPFRAC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Vestre Viken Hospital Trust (Other)
Collaborators: Oslo Metropolitan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015/2147
Record Dates: First submitted 2016-05-04; First posted 2016-05-23 (Estimated); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Femoral Neck Fractures
MeSH Terms: conditions — Femoral Neck Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional training group (Experimental): Participation in a functional training program in addition to usual care. The functional training program is initiated by the nurses and consists of walking, sit-to-stands, balance training, weight transfer training, knee squats. The program is performed 4 times a day for 3 weeks while at short-term stays.
  Interventions: Other: Functional training program
- Control group (No Intervention): Usual care only. No participation in the functional training program while at short-term stays.

INTERVENTIONS:
Other: Functional training program — Patients treated for hip fracture participate in a functional training program during their short-term stays at nursing homes. The program is initiated by the nurses 4 times a day for 3 weeks as part of the habitual routine.
  Arms: Functional training group

SUMMARY:
The survivors after hip fracture often report severe pain and loss of physical functioning. The poor outcomes cause negative impact on the person's physical functioning and quality of life and put a financial burden on society. It is important to continue and progress the functional training that already started at the hospital, while the patients are transferred to short-term stays in a nursing home before they are returning to home. The aim presently is to examine the effects of a functional training program by a RCT design, initiated by the physiotherapist and performed by the nurses, on physical functioning while the patients are at short term stays in primary health care.

DETAILED DESCRIPTION:
Functional training, such as walking and transfers, ought to be an important part of the rehabilitation after hip fracture. We have an assumption that it is of utmost importance to continue and progress the functional training that started in the acute phase at the hospital, also during the sub-acute phase while the patients are at short-term stays in nursing homes. However, there are indications of lack of resources in the nursing homes and that the nurses may be less concerned with their role and participation in the patients' rehabilitation process. Possibly, this creates a discontinuity in the rehabilitation efforts during short-term stays that may have a negative impact on the patients' recovery of physical functioning.

In this study the aim is to continue and progress the functional training started during hospital stay, such as training in walking and further on repetitive sit-to-stands, as part of the daily habitual routine during short-term stays in the nursing homes. This type of functional training may be motivational and easily recognizable to the patients, and it can also be carried out by the nursing staff with only initial guiding from a physiotherapist. There is lack of knowledge on the effect of additional functional training, incorporated as part of the habitual daily routine during short-term stays, on the patients' immediate and long term recovery of physical functioning and activity level after hip fracture, compared to usual care alone.

The study is designed as a single-blind randomized controlled trial (RCT), comparing the effects of additional functional training (functional training group)to usual care alone (control group) during short-term stays in nursing homes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an acute low-energy hip fracture (intracapsular, trochanteric or subtrochanteric) and treated surgically, ≥ 65 years of age, living in their own homes prior to the fracture, and able to give an informed consent.

Exclusion Criteria:

* Patients unable to walk 10 meters with or without a walking aid prior to the fracture, have a score of less than 15 points on Minimal Mental Status Evaluation (MMS-E) in the acute phase, have a pathological fracture, life expectancies of less than three months, medical contraindications for training, or are incapable of understanding and speaking the Norwegian language.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 140 (Actual)
Dates: Start 2016-05-30 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in the performance-based Short physical performance battery (SPPB) | Change 5 days - 3 weeks, change 5 days - 3 months, change 5 days - 12 months after surgery
  Measurement of physical functioning

SECONDARY OUTCOMES:
Change in the performance-based measure Timed Up & Go (TUG) | Change 5 days - 3 weeks, change 5 days - 3 months, change 5 days - 12 months after surgery
  Measurement of mobility
Change in the performance-based measure Hand grip strength | Change 5 days - 12 months
  Dynamometer
Descriptive performance-based measurement of physical activity, an accelerometer (activPAL) | Descriptive from day 5 to 19 after surgery
  Measurement of physical activity
Pain in rest and while walking | Change 5 days - 3 weeks, change 5 days - 3 months, change 5 days - 12 months after surgery
  Questionnaire
EuroQol (European quality of life) health status measure | Change 5 days - 3 weeks, change 5 days - 3 months, change 5 days - 12 months after surgery
  Questionnaire
University of California Los Angeles (UCLA) activity scale | Change 5 days - 3 weeks, change 5 days - 3 months, change 5 days - 12 months
  Questionnaire
New Mobility Scale (NMS) | Change 5 days - 12 months after surgery
  Questionnaire
Walking Habits | Change 5 days - 3 months, change 5 days - 12 months after surgery
  Questionnaire
Fall efficacy scale (FES) | Change 5 days - 3 weeks, change 5 days - 3 months, change 5 days - 12 months after surgery
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Kristi E Heiberg, PhD, Study Chair — Bærum Hospital Vestre Viken HF
Locations (1):
- Bærum Hospital Vestre Viken, Department of medical research, Sandvika, Drammen, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Beckmann M, Bruun-Olsen V, Pripp AH, Bergland A, Smith T, Heiberg KE. Effect of an additional health-professional-led exercise programme on clinical health outcomes after hip fracture. Physiother Res Int. 2021 Apr;26(2):e1896. doi: 10.1002/pri.1896. Epub 2021 Jan 28. PMID 33506973
- [Derived] Heiberg KE, Bruun-Olsen V, Bergland A. The effects of habitual functional training on physical functioning in patients after hip fracture: the protocol of the HIPFRAC study. BMC Geriatr. 2017 Jan 17;17(1):23. doi: 10.1186/s12877-016-0398-8. PMID 28095787